CLINICAL TRIAL: NCT06299657
Title: Project IMPROVE: Intervention for Managing Physical Reactions to Overwhelming Emotions
Brief Title: Intervention for Managing Physical Reactions to Overwhelming Emotions
Acronym: IMPROVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Nicholas Allan, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023H0286
Record Dates: First submitted 2024-03-01; First posted 2024-03-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Anxiety; Substance Use Disorders
MeSH Terms: conditions — Anxiety Disorders; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive one of two possible interventions.
Who Masked: Outcomes Assessor
Masking Description: Raters completing the outcome assessments will be blind to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IMPROVE (Experimental): In this arm, participants will receive the IMPROVE intervention, a clinician-delivered protocol targeting anxiety and uncertainty.
  Interventions: Behavioral: IMPROVE
- PHET (Active Comparator): In this arm, participants will receive a clinician-delivered protocol with a digital component, called PHET. PHET focuses on healthy living more broadly and does not include information about anxiety or uncertainty.
  Interventions: Behavioral: PHET

INTERVENTIONS:
Behavioral: IMPROVE — IMPROVE is an individual manualized intervention.
  Session1 includes:
  * psychoeducation focusing on anxiety, its role in contributing to substance use, and the maintaining role of fear of bodily sensations
  * guided discussion of maladaptive thoughts about bodily sensations related to anxiety
  * how to challenge bodily sensations cognitively
  * generating three takeaways about the benign nature of anxiety
  Session 2 includes:
  * review of homework
  * psychoeducation focusing on the role of uncertainty in anxiety and identifying how new information can inform beliefs about uncertainty.
  * when to challenge thoughts related to uncertainty and when to use acceptance regarding uncertainty.
  Session 3 includes:
  * review interoceptive exposure (IE) and behavioral exercises (BE) for progress
  * revisit beliefs related to cognitive biases
  * discuss areas where skills can be used moving forward
  Arms: IMPROVE
Behavioral: PHET — Clinicians will administer PHET using a Powerpoint presentation focused on healthy living habits, including healthy eating, water consumption, and sleep hygiene. Clinicians will guide participants through an exercise using the USDA "food tracker" to plan, record, and monitor nutritional information of meals. PHET also includes a digital program that will include EDUCATION, MY CURRENT MOOD, and BEHAVIORAL ACTIVITY tabs.
  Arms: PHET

SUMMARY:
The clinical trial aims to conduct a feasibility, acceptability, and usability clinical trial of a modular CBT-based and technologically enhanced intervention for people with an SUD and recently enrolled in IOP, probe target engagement and change in clinical outcomes, and examine attrition rates in IOP.

This study will enroll 40 adults who are currently enrolled in IOP, have a substance use disorder, and experience elevated anxiety. 20 individuals will be randomized to the experimental intervention, "Intervention for Managing Physical Reactions to Overwhelming Emotions" (IMPROVE), and 20 individuals will be randomized to the active control group, "Physical Health Education Treatment" (PHET).

Participants will be asked to complete a baseline assessment of mood, substance use, and psychophysiology. Participants will then completed ecological momentary assessments (EMA) via smartphone technology 4 times a day for ~ 28 days (the day following the baseline assessment until the 3rd intervention session). Participants will complete one 45 minute - 1 hour intervention each week for 3 weeks (either the IMPROVE or PHET intervention, pending randomization). Following the last intervention session, participants will return to the lab to complete a post-intervention assessment that mirrors the baseline assessment and then complete follow-up surveys 1- and 3-months post intervention.

DETAILED DESCRIPTION:
Substance use disorders (SUDs) represent a significant public health problem across the globe. Anxiety commonly co-occurs with SUD. This is alarming given elevated anxiety is both common and deleterious in people with an SUD and elevated anxiety significantly mitigates a person's ability to complete SUD treatment, to reduce substance use and maintain abstinence, and to maintain quality of life for those in recovery from SUD. Substance misuse and anxiety commonly co-occur due to 1) substance use to cope with anxiety symptoms, sensations, and triggers (uncertainty); and 2) heightened negative affective states that are experienced similarly across craving, withdrawal, anxiety, and stress. Intensive Outpatient Programs (IOPs) for substance use offer structured therapeutic services and support to individuals struggling with addiction, providing them with the necessary treatment and coping skills while allowing them to continue with their everyday activities. However, it has been estimated that only 50% of people who enroll in an IOP complete the program and 60% of those who do complete an IOP relapse within the first two years. Anxiety poses a significant barrier to successfully addressing substance misuse given.

In spite of this, there are no empirically supported treatments to reduce cognitive biases common to anxiety and SUDs. The investigators have iteratively developed a modular intervention rooted in cognitive behavioral therapy (CBT) called Intervention for Managing Physical Reactions to Overwhelming Emotions (IMPROVE). IMPROVE targets anxiety sensitivity (AS), or fear of anxious arousal, and intolerance of uncertainty (IU), or distress when experiencing uncertainty or ambiguity. The next step in development is a pilot acceptability, feasibility, and usability trial during which the investigators would collect preliminary effect size estimates of subjective and objective markers of AS, IU, and substance use-related outcomes. The investigators propose to conduct a randomized controlled trial comparing IMPROVE to an active control, Physical Health Education Treatment (PHET) in 40 adults enrolled in the IOP at Talbot Hall, The Ohio State University Wexner Center.

Specific Aims

Aim 1. Conduct a feasibility, acceptability, and usability clinical trial of a modular CBT-based and technologically enhanced intervention for people with an SUD and recently enrolled in IOP. Adults recently enrolled in the Talbot Hall IOP program and reporting elevated anxiety (PROMIS Anxiety Short Form total score of 13 or greater) will be randomized to IMPROVE (n = 20) or PHET (n = 20). Participants will complete a screen, multimodal assessment battery, and a week of brief surveys throughout the day via ecological momentary assessment (EMA) to capture baseline emotional distress, substance use, cravings, and withdrawal. Participants will then be randomized to a treatment arm, both of which include three weeks of face-to-face treatment supplemented by two weeks of mobile app use. Participants will complete post-intervention multimodal assessments and in-depth qualitative interviews. Finally, participants will complete the clinical assessment battery at 1- and 3-month follow-up. The investigators will assess whether IMPROVE (and PHET) meet predefined benchmarks for acceptability, feasibility, and usability.

Aim 2. Probe target engagement and change in clinical outcomes. In the context of the randomized controlled trial the investigators will: 2a) Examine whether IMPROVE reduces subjective and objective AS and IU (primary targets) and 2b) whether changes in AS and IU are associated with changes in anxiety symptoms, craving, and withdrawal sensations (primary outcomes). The investigators will also: 2c) Conduct exploratory analyses that estimate the effects of treatment-related factors (e.g., digital engagement) on changes in AS, IU, and clinical outcomes.

Aim 3. Examine attrition rates in IOP. In the context of the randomized controlled trial (RCT) the investigators will: 3a) Examine whether IMPROVE increases engagement, reduces attrition, and improves IOP completion rates.

Background & Rationale

Anxiety and SUD covary highly; further, anxiety in those with an SUD is associated with increased severity and less likelihood to remain in and benefit from SUD treatment. In our own research, the investigators have found that two transdiagnostic risk factors for anxiety are also strongly implicated in SUDs. Anxiety sensitivity, or fear of anxiety sensations, and intolerance of uncertainty, or distress experienced in the presence of uncertainty or ambiguity not only predict the etiology of anxiety and related disorders, but also predict poor substance use outcomes, including treatment dropout when enrolled in a SUD program.

The investigators have developed a modular CBT-based intervention for anxiety and related emotional distress disorders. The investigators have iteratively refined the AS and IU modules used in IMPROVE together and separately across numerous pilot trials in adults. Findings from these studies demonstrate that IMPROVE treatment components are: 1) rated as highly acceptable and feasible and 2) associated with reductions in anxiety sensitivity, intolerance of uncertainty, and emotional distress disorders. Our pilot data, which includes testing the anxiety sensitivity module in a sample of adults receiving medication-assisted therapy for an opioid use disorder (OUD), demonstrates that IMPROVE is well-positioned for adaptation as a supplemental treatment for individuals enrolled in an IOP.

ELIGIBILITY:
Inclusionary Criteria:

Participants will be eligible for enrollment if they:

1. recently enrolled in the Talbot Hall IOP
2. >18 years old
3. PROMIS Anxiety Short Form total score is 13 or greater

Exclusionary Criteria:

1. do not pass the Informed Decision-Making Capacity (IDMC) screener, suggesting severe cognitive impairment
2. presence of a psychiatric or medical condition that would prevent them from providing informed consent or from participating in the treatments (e.g., psychosis, mania, acute intoxication)
3. no or limited access to a smartphone that is compatible with the EMA application

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Intolerance of Uncertainty-12 Scale | Change will be assessed from baseline to the post-intervention session, occurring four weeks after the baseline session
  Intolerance of uncertainty is measured using the 12-item Intolerance of Uncertainty Scale - Short Form. Each item is measured on a 5-point scale from (1) Not At All Characteristic Of Me to (5) Entirely Characteristic Of Me. Higher scores indicate worse intolerance of uncertainty with scores ranging from 12 to 60.
Anxiety Sensitivity-3 Scale | Change will be assessed from baseline to the post-intervention session, occurring four weeks after the baseline session
  Anxiety sensitivity is measured using the 18-item Anxiety Sensitivity Scale. Each item is measured on a 5-point scale from (1) Very Little to (5) Very Much. Higher scores indicate higher anxiety sensitivity with scores ranging from 18 to 90.
PROMIS Anxiety Short Form | Change will be assessed from baseline to a) 1-month follow-up and b) 3-month follow-up
  Anxiety symptoms are measured using the 8-item PROMIS Anxiety Short Form. Each item is measured on a 5-point scale from (1) Never to (5) Always. Higher scores indicate increased anxiety symptoms with scores ranging from 8 to 40.
Timeline Followback | Change will be assessed from baseline to a) 1-month follow-up and b) 3-month follow-up
  Substance use is measured using The Timeline Followback (TLFB). The TLFB asks participants to estimate their substance use 7 days to 2 years prior to the interview date.
Desire for Drug Questionnaire | Change will be assessed from baseline to a) 1-month follow-up and b) 3-month follow-up
  Craving for opioids will be measured using the 13-item Desire for Drug Questionnaire. Each item is measured on a 7-point scale from (1) Strongly Disagree to (7) Strongly Agree. High scores indicate increased craving with scores ranging from 13 to 91.
Penn Alcohol Craving Scale | Change will be assessed from baseline to a) 1-month follow-up and b) 3-month follow-up
  Craving for alcohol will be measured using the 5-item Penn Alcohol Craving Scale. Each item is measured on a 7-point scale from 0 to 6. High scores indicate increased craving with scores ranging from 0 to 30.
Hyperkatifeia Interference Scale - Alcohol Version. | Change will be assessed from baseline to a) 1-month follow-up and b) 3-month follow-up
  Withdrawal symptoms for alcohol will be measured using the 7-item Hyperkatifeia Interference Scale - Alcohol Version. Each item is measured on a sliding scale from (0) Did Not Interfere to (100) Completely Interfered. High scores indicated higher interference.
Clinical Institute Withdrawal Assessment Alcohol Scale Revised. | Change will be assessed from baseline to a) 1-month follow-up and b) 3-month follow-up
  Withdrawal symptoms for alcohol will be measured using the clinician-administered Clinical Institute Withdrawal Assessment Alcohol Scale Revised. The measure includes heart rate and blood pressure readings followed by 10 items. Each item is measured on an 8-point scale from 0 to 7.
Hyperkatifeia Interference Scale - Opioid Version. | Change will be assessed from baseline to a) 1-month follow-up and b) 3-month follow-up
  Withdrawal symptoms for opioids will be measured using the 7-item Hyperkatifeia Interference Scale - Opioid Version. Each item is measured on a sliding scale from (0) Did Not Interfere to (100) Completely Interfered. High scores indicated higher interference.
Subjective Opiate Withdrawal Scale | Change will be assessed from baseline to a) 1-month follow-up and b) 3-month follow-up
  Withdrawal symptoms for opioids will be measured using the 16-item Subjective Opiate Withdrawal Scale. Each item is measured on 5-point scale from (0) Not At All to (4) Extremely. High scores indicate increased withdrawal symptoms.
NPU Threat Task | Change will be assessed from baseline to the post-intervention session, occurring four weeks after the baseline session
  Intolerance of uncertainty will be measured using the NPU Threat Task. The task includes a brief, mild electric shock to elicit aversive responding. The task will be a modified version of Grillon and colleagues' No-, Predictable-, Unpredictable -Threat (NPU) startle paradigm11. The NPU-Threat task includes three within-subjects conditions - no shock (N), predictable shock (P), and unpredictable shock (U). Total task time is around 13 minutes.
Straw Breathing Avoidance Task | Change will be assessed from baseline to the post-intervention session, occurring four weeks after the baseline session
  Anxiety sensitivity will be measured using the Straw Breathing Avoidance Task. The Straw Breathing Avoidance Task (SB-BAT) is a behavioral task that is used as an index of anxiety sensitivity. The SB-BAT reliably produces bodily sensations mimicking those induced by anxiety by breathing through a coffee straw for two minutes at a rate of 30 breaths per minute, guided by an audio recording. Individuals rate their reaction to that arousal in real-time via self-report ratings, ranging from 0 (no fear) to 100 (extreme fear or panic).
Emotion Picture Paradigm Task | Change will be assessed from baseline to the post-intervention session, occurring four weeks after the baseline session
  Neural responses of anxiety sensitivity will be measured using the Emotion Picture Paradigm Task. Individual differences in AS will be assessed using a modified version of the emotion picture paradigm (EPP) during continuous electroencephalography (EEG) recording. The task is uniquely designed to capture neural reactivity to anxiety sensitivity (AS) stimuli. Participants will observe 80 images in four categories: unpleasant, pleasant, neutral, and AS. Images will be presented for 6 seconds, in blocks of 10 images. Blocks of each picture type are presented twice (20 images/type).

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University Department of Psychiatry and Behavioral Health, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified demographic and clinical data collected as part of this project will be available as raw individual level data for sharing with external researchers working at an institution with a Federalwide Assurance (FWA) for the Protection of Human Subjects. Data will therefore be available for secondary analytic purposes. Names and institutions of persons either given or denied access to data will be tracked by our Administrative Core and will be available upon request from the sponsor. Data will not be available for data sharing until after this project is complete and the primary outcomes are published.
Supporting Information: Study Protocol
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for at least the next two years. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial individual participant data (IPD) can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).